CLINICAL TRIAL: NCT03188510
Title: Relative Bioavailability of LY3074828 Solution Formulation in Pre-Filled Syringes Compared to Lyophilized Formulation After Single Subcutaneous Administration
Brief Title: A Study of Two Different Formulations of LY3074828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16455; I6T-MC-AMAE (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reference: 250 mg LY3074828 (Experimental): 250 mg LY3074828 lyophilized formulation administered subcutaneously (SC) as 3 injections
  Interventions: Biological: LY3074828
- Test 1: 250 mg LY3074828 (Experimental): 250 mg LY3074828 solution formulation administered as SC injections in two prefilled syringes
  Interventions: Biological: LY3074828
- Test 2: 500 mg LY3074828 (Experimental): 500 mg LY3074828 solution formulation administered as SC injections in four prefilled syringes
  Interventions: Biological: LY3074828

INTERVENTIONS:
Biological: LY3074828 — Administered SC

SUMMARY:
The purpose of this study is to look at the amount of the study drug, LY3074828, that gets into the blood stream and how long it takes the body to get rid of LY3074828 when given as different formulations. The tolerability of LY3074828 will also be evaluated and information about any side effects experienced will be collected.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be approximately 13 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 1 month of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have significant allergies to humanised monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or sever post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reference: 250 mg LY3074828: Participants received 250 mg LY3074828 lyophilized formulation, as 3 subcutaneous (SC) injections.
- Test 1: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation in 2 prefilled syringes (PFSs), as SC injections.
- Test 2: 500 mg LY3074828: Participants received 500 mg LY3074828 solution formulation in 4 PFSs, as SC injections.
Period: Overall Study
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828
Started | 18 | 18 | 18
Received at Least 1 Dose of Study Drug | 18 | 18 | 18
Completed | 18 | 17 | 18
Not Completed | 0 | 1 | 0
Not completed — Inappropriate behavior with site staff | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Reference: 250 mg LY3074828: Participants received 250 mg LY3074828 lyophilized formulation, as 3 SC injections
- Test 1: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation in 2 PFSs, as SC injections
- Total: Total of all reporting groups
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828 | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (12.6) | 42.1 (11.0) | 42.5 (10.3) | 42.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 8 | 26
  Male | 8 | 10 | 10 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 6 | 14
  Not Hispanic or Latino | 14 | 14 | 12 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 7 | 26
  White | 9 | 8 | 9 | 26
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Dose-normalized Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (DN-AUC[0-tlast]) of LY3074828
Description: PK: Dose-normalized Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (DN-AUC[0-tlast]) of LY3074828 was evaluated. Unit of measure expansion: microgram*day per milliliter per milligram (µg*day/mL/mg).
Time Frame: Predose; 2, 6, 24, 72, 168, 240, 336, 504, 672, 1008, 1344, 1680 and 2016 hours postdose
Population: All enrolled participants who received at least one dose of LY3074828 and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*day/mL/mg
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828
Number analyzed (Participants) | 18 | 17 | 18
µg*day/mL/mg | 1.06 (27) | 1.03 (40) | 1.04 (32)
Statistical Analysis 1: Comparison: Reference: 250 mg LY3074828 vs Test 1: 250 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 0.971, 90% CI 2-sided [0.805 to 1.17]
Statistical Analysis 2: Comparison: Test 1: 250 mg LY3074828 vs Test 2: 500 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 1.01, 90% CI 2-sided [0.841 to 1.22]
Statistical Analysis 3: Comparison: Reference: 250 mg LY3074828 vs Test 2: 500 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 0.985, 90% CI 2-sided [0.819 to 1.18]

2. Primary Outcome: PK: Dose-normalized Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (DN-AUC[0-∞]) of LY3074828
Description: PK: Dose-normalized Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (DN-AUC[0-∞]) of LY3074828 was evaluated.
Time Frame: Predose; 2, 6, 24, 72, 168, 240, 336, 504, 672, 1008, 1344, 1680 and 2016 hours postdose
Population: All enrolled participants who received at least one dose of LY3074828 and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg.day/mL/mg
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828
Number analyzed (Participants) | 18 | 17 | 18
µg.day/mL/mg | 1.07 (27) | 1.05 (40) | 1.05 (32)
Statistical Analysis 1: Comparison: Reference: 250 mg LY3074828 vs Test 1: 250 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 0.978, 90% CI 2-sided [0.811 to 1.18]
Statistical Analysis 2: Comparison: Test 1: 250 mg LY3074828 vs Test 2: 500 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 1.00, 90% CI 2-sided [0.833 to 1.21]
Statistical Analysis 3: Comparison: Reference: 250 mg LY3074828 vs Test 2: 500 mg LY3074828; Test type: Other; Ratio of geometric least squares means = 0.982, 90% CI 2-sided [0.817 to 1.18]

3. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (TE-ADA)
Description: Number of participants with positive treatment emergent anti-drug antibodies was summarized by treatment group. A treatment-emergent ADA (TEADA) was defined as: having a negative ADA at baseline and an ADA titer greater than or equal to 1:20 (that is (i.e.), greater than 2-fold from the minimal required dilution of 1:10) any time post baseline (i.e., treatment-induced); or a 4-fold or greater change in ADA titer from baseline for participants that had a detectable ADA titer at baseline (i.e., treatment boosted).
Time Frame: Predose Day 1 Through Day 85
Population: All randomized participants who received at least one dose of LY3074828 and had evaluable anti-drug antibody measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828
Number analyzed (Participants) | 18 | 17 | 18
Participants | 7 | 6 | 7

ADVERSE EVENTS:
Time Frame: Up to 85 days after administration of study drug
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | Reference: 250 mg LY3074828 | Test 1: 250 mg LY3074828 | Test 2: 500 mg LY3074828
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 16/18 | 15/18 | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference: 250 mg LY3074828 (N=18) | Test 1: 250 mg LY3074828 (N=18) | Test 2: 500 mg LY3074828 (N=18)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 3 (4) | 1 (1) | 3 (3)
Injection site reaction (General disorders) | 15 (32) | 15 (24) | 18 (55)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-04-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03188510/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT03188510/SAP_001.pdf